CLINICAL TRIAL: NCT02008669
Title: Evaluation of the Nutritional Status of Patients With Multiple Sclerosis and Relationship With Fatigue
Brief Title: Evaluation of Nutritional Status and Fatigue in Patients With Multiple Sclerosis
Acronym: NUTRISEP
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0022
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, Fatigue, Nutritional Status, Disability.
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological analysis in serum: magnesium, albumin, Vitamin B12, Vitamin D, Calcium, Iron.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Sclerosis cases: All patients will undergo the following interventions
  * Gustatory sensitivity test using Taste strips
  * Blood sampling
  * Questionnaires
  Interventions: Procedure: Blood sampling; Other: Gustatory sensitivity test using Taste strips; Other: Questionnaires

INTERVENTIONS:
Procedure: Blood sampling — A blood sample will be taken from each patient and the following parameters will be assessed : magnesium, albumin, Vitamin B12, Vitamin D, Calcium, Iron.
Other: Gustatory sensitivity test using Taste strips — 16 Taste Strips impregnated with 4 flavors (sweet, sour, salty, bitter, each flavor present at 4 different concentrations), are offered to the patient one after the other in a so-called pseudorandomized sequence. The task of the patient is to choose one of the following answers: sweet / sour / salty / bitter / no taste.
  Each correct answer is granted one point. In addition to the impregnated strips, two tasteless strips can be integrated in the examination at any point of time (no point)
Other: Questionnaires — Evaluation of the following parameters by validated questionnaires (name of the questionnaire in bracket):
  * Fatigue (EMIF-SEP)
  * Dysphagia (DYMUS)
  * Food intake (semi-structured questionnaire)
  * Depression (BDI-II)
  * Daily energy expenditure (NAP)
  * Visual analog scale to study quality of sleep

SUMMARY:
Multiple sclerosis (MS) is a chronic progressive neurological disease, the leading cause of disability after injury accidents in young adults. Among the many symptoms, fatigue is very common with a significant impact on quality of life. Also, the disability caused by multiple sclerosis can alter food intake and can cause nutritional deficiencies. Nutrients such as proteins, minerals (iron, calcium, magnesium), some vitamins (B12, 25 OHD) are often deficient in this population with consequences in physical performance such as endurance and muscle strength. We propose to study the link between fatigue and shortcomings encountered in a defined population of MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old
* Expended disability status scale (EDSS) between 0 and 7
* Diagnosis of MS according to the revised criteria of McDonald
* Clinically stable patients in the past 3 months
* Coverage of the social insurance
* Informed consent to participate

Exclusion Criteria:

* Cognitive disorders that can hinder answering questionnaires
* Presence of uncontrolled metabolic disease(s)
* Malabsorption
* Patients with a gastrostomy
* Active cancer under treatment
* Anorexia
* Pregnancy or breast feeding
* Severe psychiatric disorder(s)
* No informed consent to participate
* No coverage by the social insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS defined according to the revised diagnostic criteria of Mac Donald, with ages between 18 to 65 years with an Expended disability status scale (EDSS) between 0 and 7 and followed in the services of neurology or physical medicine and rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Correlation between the score of fatigue EMIF-SEP and the dosage of nutrients in blood (vitamins, minerals, proteins) adjusted by the EDSS status | Baseline
  The objective is to construct and validate a regression model between the scale of fatigue and biological variables

SECONDARY OUTCOMES:
Presence or absence of sociodemographic variables | Baseline
Presence or absence of clinical manifestations | Baseline
Level of physical activity and daily energy expenditure | Baseline
Assessment of dysphagia according to the score of the Dymus Test | Baseline
Score of the taste sensibility test | Baseline
Score of the Beck depression inventory test | Baseline
  This test is a 21-question multiple-choice self-report inventory for measuring the severity of depression
Score of the visual analog scale for the evaluation of sleep quality | Baseline
Score of the Nutrition and Eating Habits Questionnaire | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Donzé, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (12):
- France (12):
  - Centre Hospitalier Universitaire de Caen, Caen, Basse-Normandie
  - Centre Hospitalier d'Arras, Arras, Hauts-de-France
  - Centre Hospitalier de Boulogne, Hôpital Duchenne, Boulogne-sur-Mer, Hauts-de-France
  - Centre Hospitalier de Calais, Calais, Hauts-de-France
  - Centre Hospitalier de Douai, Douai, Hauts-de-France
  - Groupement des Hôpitaux de l'Institut Catholique de Lille, Lille, Hauts-de-France
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Hauts-de-France
  - Centre Hospitalier de Sambre-Avenois, Maubeuge, Hauts-de-France
  - Centre Hélène Borel, Raimbeaucourt, Hauts-de-France
  - Centre Hospitalier Dron de Tourcoing, Tourcoing, Hauts-de-France
  - Centre Hospitalier de Valenciennes, Valenciennes, Hauts-de-France
  - Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie